CLINICAL TRIAL: NCT01735916
Title: MIRACLE EF Clinical Study
Acronym: MIRACLE EF
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was terminated early due to low enrollment.
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MIRACLE EF
Record Dates: First submitted 2012-11-15; First posted 2012-11-28 (Estimated); Results first posted 2014-10-06 (Estimated); Last update posted 2017-11-06 (Actual); Status verified 2017-10

CONDITIONS: Congestive Heart Failure; Left Bundle Branch Block; Systolic Heart Failure
MeSH Terms: conditions — Heart Failure; Bundle-Branch Block; Heart Failure, Systolic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CRT-P ON (Active Comparator): CRT-P Implant CRT-P ON
  Interventions: Device: CRT-P Implant
- CRT-P OFF (Placebo Comparator): CRT-P Implant CRT-P OFF
  Interventions: Device: CRT-P Implant; Device: CRT-P OFF

INTERVENTIONS:
Device: CRT-P Implant — The Medtronic Consulta CRT-P (models C3TR01, C4TR011) dual chamber implantable pacemaker with cardiac resynchronization therapy (CRT-P) is a multi-programmable cardiac device that monitors and regulates the patient's heart rate by providing single or dual chamber rate-responsive bradycardia pacing, and sequential biventricular pacing.
  The device senses the electrical activity of the patient's heart using the electrodes of the implanted atrial and right ventricular leads. It then analyzes the heart rhythm based on selectable detection parameters. The device responds to bradyarrhythmias by providing bradycardia pacing therapy.
  Simultaneous or sequential biventricular pacing is used to provide patients with cardiac resynchronization therapy. The device also provides diagnostic and monitoring information that assists with system evaluation and patient care.
  Other Names: Cardiac Resynchronization Therapy Pacemaker (CRT-P); Consulta CRT-P; C4TR01
Device: CRT-P OFF — Device programmed to minimal pacing at 40 beats/minute. Device and arrhythmia diagnostics may remain enabled.
  Arms: CRT-P OFF

SUMMARY:
This study is looking at whether the electrical treatment provided by a special type of pacemaker called a Cardiac Resynchronization Therapy (CRT) pacemaker may keep a patient's heart failure from getting worse. When the lower heart chambers (i.e. ventricles) are electrically paced to beat together by the CRT pacemaker, blood may be pumped to the body more efficiently.

The CRT pacemaker being studied in this clinical trial is approved by the US Food and Drug Administration (FDA) for patients with moderate to severe heart failure, whose hearts pump blood inefficiently. In the MIRACLE EF study, patients who have heart failure with slightly less inefficient hearts will be observed to see if the electrical pacing treatment is better than not getting the treatment. This study is being conducted to support FDA approval of this type of pacemaker for people whose heart failure is less inefficient.

DETAILED DESCRIPTION:
Medtronic, Inc. is sponsoring the MIRACLE EF study, a prospective, randomized, controlled, double-blinded, global multi-center, Cardiac Resynchronization Therapy (CRT) in Heart Failure (HF) clinical study. The purpose of this study is to evaluate market released CRT pacemaker (CRT-P) devices in symptomatic HF patients with less severe left ventricular systolic dysfunction, specifically patients with reduced left ventricular ejection fraction (LVEF) in the range of 36% to 50%. This study will support expansion of indications for CRT worldwide. The outcome of this study is expected to support modification of existing U.S. and Japanese labeling for Medtronic's implantable CRT-P devices and to provide further evidence to support changes to cardiology practice guidelines (ACC/AHA, ESC guidelines) regarding the use of CRT in patients with mild to moderate HF.

Following enrollment and the baseline assessment, eligible subjects will be implanted with a CRT-P system and randomized in a 2:1 fashion to either treatment (CRT-P ON) or control (CRT-P OFF) groups. Study subjects will be followed for a minimum of 24 months or until study closure, and will remain in their randomized groups until their 60 month visit or until the study is stopped, whichever comes first. The effectiveness of CRT-P in this population will be assessed using a composite endpoint of time to first event, with event defined as All-cause mortality or HF Event. To assess the safety of CRT-P in this population, the primary safety endpoint will measure freedom from system-related complications at 6 months post-implant.

ELIGIBILITY:
Inclusion Criteria:

* Patient has diagnosis of chronic heart failure > 90 days in duration
* Has left ventricular ejection fraction (LVEF) between 36% and 50%, inclusive, as documented at baseline or within 30 days prior to enrollment
* Is either: (a) NYHA Class III at enrollment or at baseline OR (b) NYHA Class II at enrollment or at baseline, with a documented hospitalization for HF in the 12 months prior to enrollment OR (c) NYHA Class II at enrollment or at baseline, without a documented hospitalization for HF in the prior 12 months, but with BNP ≥250 pg/ml or NT-proBNP ≥1000 pg/ml
* Has documented left bundle branch block (LBBB) with QRS ≥130ms at baseline or within 30 days prior to enrollment.
* Is in sinus rhythm at time of enrollment or at the baseline visit.
* Has had no additions to or subtractions from non-diuretic heart failure medical therapy within 30 days prior to enrollment
* Is on maximum tolerated (guideline) dosages of medications in ACC/AHA guidelines for HF, Ischemic Heart Disease, Hypertension and AF as appropriate.
* Has signed and dated the study informed consent.
* Is able to receive a pectoral CRT-P implant.
* Is expected to remain available for follow-up visits.
* Is willing and able to comply with the Clinical Investigation Plan.

Exclusion Criteria:

* Requires permanent cardiac pacing.
* Indicated for implantable cardioverter defibrillator (ICD), such as for secondary prevention of prior sudden cardiac arrest, related to prior history of ventricular tachycardia and/or ventricular fibrillation.
* Less than 18 years of age, or under a higher minimum age requirement as defined by local law.
* Unstable angina or an acute MI within 40 days prior to enrollment.
* Coronary artery bypass graft (CABG) or percutaneous coronary intervention (PCI) within the 90 days prior to enrollment.
* Chronic (permanent) atrial arrhythmias. Chronic (permanent) atrial arrhythmias are defined as cases of long-standing atrial fibrillation (e.g., greater than 1 year) in which cardioversion has not been indicated or attempted.
* Cardioversion for atrial fibrillation within 30 days prior to enrollment.
* Treatable pericardial constraint within 30 days prior to enrollment.
* Restrictive (infiltrative) cardiomyopathies, such as amyloidosis, sarcoidosis, or hemochromatosis.
* Enrolled in a concurrent study, with the exception of a study-manager approved study that is strictly observational in nature and does not confound the results of this study (e.g. registries).
* Life expectancy of less than 24 months due to non-cardiac conditions.
* Pregnant, or of childbearing potential and not on a reliable form of birth control.
* CRT-P, pacemaker, ICD or CRT-D device implanted previously, or currently.
* Restrictive, hypertrophic, or reversible cardiomyopathy.
* Mechanical right heart valve.
* Primary valvular disease and is indicated for valve repair or replacement.
* Heart transplant, or is currently on a heart transplant list.
* Significant renal dysfunction, as manifested by serum creatinine level >2.5 mg/dl or ≥275 μmol/L or estimated glomerular filtration rate (GFR) ≤30 mL/min/1.73 m2, which is documented within the 30 days prior to enrollment or at baseline.
* Significant hepatic dysfunction, as evidenced by a hepatic function panel (serum) > 3 times upper limit of normal, which is documented within the 30 days prior to enrollment or at baseline.
* Chronic or treatment-resistant severe anemia (hemoglobin <10.0 g/dL), which is documented within the 30 days prior to enrollment or at baseline.
* On intravenous inotropic drug therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2012-12; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cecilia Linde, MD PhD, Study Chair — Karolinska University Hospital
Locations (73):
- United States (69):
  - John Muir Medical Center, Cor Cardiovascular Specialists, John Muir Medical Center (Concord), John Muir Cardiovascular Institute, Contra Costa Cardiology, Concord, California
  - Scripps Clinic Torrey Pines, Scripps Green Hospital, La Jolla, California
  - VA Greater Los Angeles Healthcare System, Los Angeles, California
  - Eisenhower Desert Cardiology Center, Eisenhower Medical Center Hospital, Rancho Mirage, California
  - Los Robles Medical Center, Thousand Oaks, California
  - Colorado Health Medical Group, Memorial Hospital Colorado Springs, Colorado Springs, Colorado
  - Hartford Hospital, Hartford, Connecticut
  - Bradenton Cardiology, Manatee Memorial Hospital, Bradenton, Florida
  - Melbourne Internal Medicine Associates / Century Research Associates, Holmes Regional Medical Center Hospital, Melbourne, Florida
  - Aventura Hospital and Medical Center, Hospital Corporation of America (Aventura), Hospital Corporation of America (Miami), Miami, Florida
  - Emory University Hospital Midtown, Atlanta, Georgia
  - WellStar Cobb Hospital, WellStar Kennestone Hospital, Marietta, Georgia
  - Advocate Medical Group, Midwest Heart Specialists (Elmhurst), Elmhurst Memorial Hospital, Elmhurst, Illinois
  - Advocate Christ Medical Center, Oak Lawn, Illinois
  - Prairie Education and Research Cooperative (Springfield IL), Prairie Education Research Consultants, St. John's Hospital (Springfield IL), Springfield, Illinois
  - McFarland Clinic PC, Ames, Iowa
  - Cardiovascular Medicine PC (Davenport IA), Trinity (Rock Island), Midwest Cardiovascular Research Foundation, Trinity Bettendorf Hospital, Davenport, Iowa
  - Midwest Cardiology Associates PA, Menorah Medical Center, Centerpoint Medical Center, Overland Park Regional Medical Center Hospital, Overland Park, Kansas
  - Lahey Hospital & Medical Center, Burlington, Massachusetts
  - Sparrow Clinical Research Institute, McLaren Hospital, Lansing, Michigan
  - William Beaumont Hospital, Royal Oak, Michigan
  - HealthEast HeartCare Clinic at Saint John's, Maplewood, Minnesota
  - Minneapolis Heart Institute Foundation, Minneapolis, Minnesota
  - The Cardiovascular Center, University of Minnesota Medical Center Fairview, Minneapolis, Minnesota
  - North Memorial Heart and Vascular Institute, North Memorial Medical Center, Robbinsdale, Minnesota
  - CentraCare Heart & Vascular Center, Saint Cloud, Minnesota
  - Minneapolis Heart Institute Foundation, Mercy Hospital (Coon Rapids MN), Unity Hospital, United Hospital, Abbott Northwestern Hospital, Saint Paul, Minnesota
  - Missouri Cardiovascular Specialists, Boone Hospital Center, Columbia, Missouri
  - Cardiovascular Consultants, P.C., Saint Luke's Hospital, Mid America Heart Institute (MAHI), Kansas City, Missouri
  - Mercy Heart and Vascular Clinic, Mercy Hospital St. Louis, St Louis, Missouri
  - Glacier View Research Institute Cardiology, Duplicate Glacier View Research Institute Hospital, Kalispell, Montana
  - Hackensack University Medical Center, Hackensack, New Jersey
  - New Mexico Heart Institute PA, Albuquerque, New Mexico
  - Buffalo Heart Group LLP, Buffalo Heart Group LLC-Cheektowaga, Mercy Hospital of Buffalo, Buffalo, New York
  - Stony Brook Islandia Clinic, Stony Brook Hauppauge, Stony Brook University Medical Center, Stony Brook, New York
  - Duke University Medical Center (DUMC), Durham, North Carolina
  - Durham VA Medical Center, Duke University Medical Center, Durham, North Carolina
  - FirstHealth Cardiology Services, FirstHealth Moore Regional Hospital, Pinehurst, North Carolina
  - Forsyth Medical Center, Novant Clinical Research Institute, Winston-Salem, North Carolina
  - Sanford Medical Center, Fargo, North Dakota
  - Lindner Research Center, The Christ Hospital, Cincinnati, Ohio
  - Ohio State University, Ohio State University Medical Center The Richard M Ross Heart Hospital, Columbus, Ohio
  - Mercy Hospital Fairfield, Mercy Hospital Anderson, The Jewish Hospital, Fairfield, Ohio
  - Integris Baptist Medical Center, Oklahoma City, Oklahoma
  - Samaritan Health Services, Corvallis, Oregon
  - Oregon Health & Science University, Portland, Oregon
  - Lehigh Valley Hospital, Allentown, Pennsylvania
  - Mercer Bucks Cardiology, Saint Mary Medical Center, Arrhythmia Institute Hospital, Newtown, Pennsylvania
  - University of Pittsburgh Medical Center UPMC Presbyterian, Pittsburgh, Pennsylvania
  - Cardiac Diagnostic Associates, York Hospital, York, Pennsylvania
  - Pee Dee Cardiology, McLeod Regional Medical Center, Florence, South Carolina
  - Arrhythmia Consultants (Greenville SC), Greenville Memorial Hospital, Greenville, South Carolina
  - Cardiology Consultants PA, Spartanburg Regional Hospital, Spartanburg, South Carolina
  - Wellmont CVA Heart Institute, Wellmont Holston Valley Medical Center, Kingsport, Tennessee
  - Centennial Heart Cardiovascular Consultants LLC, Nashville, Tennessee
  - Saint Thomas Research Institute LLC, Baptist Hospital, Nashville, Tennessee
  - Amarillo Heart Group, Northwest Texas Hospital, Amarillo, Texas
  - Cardiology Center of Amarillo, Northwest Texas Hospital, Amarillo, Texas
  - HeartPlace Cardiology Research, Baylor Heart & Vascular Hospital, Dallas, Texas
  - Methodist DeBakey Cardiology Associates, The Methodist Hospital, Houston, Texas
  - Baylor Research Institute (Plano TX), Legacy Heart Center, Plano, Texas
  - Scott & White Hospital, Temple, Texas
  - Fletcher Allen Medical Center, Burlington, Vermont
  - University of Virginia (UVA) Medical Center, Charlottesville, Virginia
  - Centra Medical Group Stroobants Cardiovascular Center, Centra Lynchburg General Hospital, Lynchburg, Virginia
  - Richmond Cardiology Associates, Bon Secours Memorial Regional Medical Center, Mechanicsville, Virginia
  - Sentara Cardiovascular Specialist, Sentara Williamsburg Regional Medical Center, Sentara Norfolk General Hospital, Sentara Virginia Beach General Hospital, Norfolk, Virginia
  - Harborview Medical Center, University of Washington (UW) Medical Center, Seattle, Washington
  - Aurora Cardiovascular Services, Aurora Sinai Medical Center, Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
- Medanta-The Medicity, Haryāna, India
- Tyumen Cardiology Center, Tyumen, Russia
- Karolinska University Hospital, Stockholm, Sweden
- University Hospitals of Birmingham NHS Foundation Trust - Queen Elizabeth Hospital, Birmingham, United Kingdom

RESULTS

PARTICIPANT FLOW:
Groups:
- No Implant Attempt: Subjects who did not undergo an implant attempt of a CRT-P device and were not randomized.
- CRT-P ON: Subjects who were implanted with a CRT-P device and device programmed to provide simultaneous or sequential biventricular pacing to provide patients with cardiac resynchronization therapy. The device also provides diagnostic and monitoring information that assists with system evaluation and patient care.
- CRT-P OFF: Subjects who were implanted with a CRT-P device and device programmed to minimal right ventricular-only pacing at 40 beats/minute. Device and arrhythmia diagnostics may remain enabled.
Period: Overall Study
Arm/Group | No Implant Attempt | CRT-P ON | CRT-P OFF
Started | 18 | 19 | 7
Completed | 0 | 0 (Study was cancelled before any subjects completed 24 months of follow-up or met any study endpoints.) | 0 (Study was cancelled before any subjects completed 24 months of follow-up or met any study endpoints.)
Not Completed | 18 | 19 | 7
Not completed — Subject not eligible to be randomized | 11 | 0 | 0
Not completed — Early termination of study by sponsor | 4 | 19 | 7
Not completed — Withdrawal by Subject | 3 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | No Implant Attempt | CRT-P ON | CRT-P OFF | Total
Number analyzed (Participants) | 18 | 19 | 7 | 44
Age, Continuous [Mean (Standard Deviation); unit: years] — Not all data were available for non-randomized subjects due to exiting prior to randomization. Age was available for 8 of the non-randomized subjects and was not available for 10 of the 18 non-randomized subjects.
  years | 68.5 (10.4) | 69.2 (10.3) | 69.3 (7.0) | 69.0 (9.5)
Sex/Gender, Customized [Number; unit: participants]
  Male | 5 | 5 | 6 | 16
  Female | 3 | 14 | 1 | 18
  Not Reported | 10 | 0 | 0 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 2 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 6 | 17 | 7 | 30
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 11 | 0 | 0 | 11
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilogram/(meter*meter)] — Not all data were available for non-randomized subjects due to exiting prior to randomization. BMI was available for 8 of the non-randomized subjects and was not available for 10 of the 18 non-randomized subjects.
  kilogram/(meter*meter) | 29.3 (4.9) | 31.5 (7.0) | 32.5 (3.6) | 31.2 (6.0)
Heart rate [Mean (Standard Deviation); unit: intrinsic beats/minute] — Not all data were available for non-randomized subjects due to exiting prior to randomization. Heart rate was available for 8 of the non-randomized subjects and was not available for 10 of the 18 non-randomized subjects.
  intrinsic beats/minute | 63.4 (12.8) | 72.6 (10.3) | 64.3 (6.7) | 68.7 (11.0)
Systolic blood pressure [Mean (Standard Deviation); unit: mm Hg] — Not all data were available for non-randomized subjects due to exiting prior to randomization. Systolic blood pressure was available for 8 of the non-randomized subjects and was not available for 10 of the 18 non-randomized subjects.
  mm Hg | 130.9 (20.7) | 131.5 (21.4) | 121.1 (19.0) | 129.2 (20.6)
Diastolic blood pressure [Mean (Standard Deviation); unit: mm Hg] — Not all data were available for non-randomized subjects due to exiting prior to randomization. Diastolic blood pressure was available for 8 of the non-randomized subjects and was not available for 10 of the 18 non-randomized subjects.
  mm Hg | 74.4 (9.4) | 74.4 (10.2) | 66.6 (11.5) | 72.8 (10.5)
New York Heart Association classification [Number; unit: participants] — New York Heart Association Classification is a measure of the degree of heart failure a subject has on a 4 class scale, with NYHA Class I being the healthiest score and NYHA Class IV being the sickest score.
  participants
    NYHA Class II | 11 | 2 | 3 | 16
    NYHA Class III | 5 | 17 | 4 | 26
    Not Reported | 2 | 0 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Mortality or Heart Failure Morbidity
Description: Primary Efficacy Endpoint: The time to first event, with event defined as:
  * All-cause mortality, or
  * HF Event, defined as either:
  * Inpatient hospitalization for HF, or
  * Outpatient event requiring invasive clinical intervention and management for HF (i.e. IV diuretics, ultrafiltration, or equivalent) and overnight stay
  Note: No endpoints were reached, so this objective was not analyzed
Time Frame: From date of randomization to date of event, assessed for a minimum of 24 months and up to 60 months
Arm/Group | CRT-P ON | CRT-P OFF
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: System-related Complication
Description: Primary Safety Endpoint: Time to first system-related complication in subjects with a successful implant.
  Note: Because of the small number of subjects, number of complications was noted between arms and a time to event analysis was not performed.
  Complication is defined as: An adverse event that results in death, involves any termination of significant device function, or requires an invasive intervention
Time Frame: From the date of implant to the date of 6 month follow-up visit
Measure: Number; unit: Complications
Arm/Group | CRT-P ON | CRT-P OFF
Number analyzed (Participants) | 19 | 7
Complications | 1 | 2

3. Secondary Outcome: Mortality
Description: Time to death between the study groups
  Note: No endpoints were reached, so this objective was not analyzed
Time Frame: From date of randomization to date of death, for a minimum of 24 months and up to 60 months
Arm/Group | CRT-P ON | CRT-P OFF
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Mortality or Heart Failure Morbidity or Worsening Systolic Function
Description: Secondary Composite Efficacy Endpoint: The time to first event, with event defined as:
  * All-cause mortality
  * HF Event, defined as either:
  * Inpatient hospitalization for HF, or
  * Outpatient event requiring invasive clinical intervention and management for HF (i.e. IV diuretics, ultrafiltration, or equivalent) and overnight stay, or
  * Worsening systolic function meeting an ICD/CRT-D indication, defined as:
  * A drop in LVEF to 35% or below, with an absolute decrease of greater than or equal to 10%, after maximum tolerated doses of guideline HF medications have been established
  Note: No endpoints were reached, so this objective was not analyzed
Time Frame: From date of randomization to date of event, assessed for a minimum of 24 months and up to 60 months
Arm/Group | CRT-P ON | CRT-P OFF
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Recurrent HF Events
Description: The frequency of HF events between the study groups
  Note: No endpoints were reached, so this objective was not analyzed
  - HF Event, defined as either:
  * Inpatient hospitalization for HF, or
  * Outpatient event requiring invasive clinical intervention and management for HF (i.e. IV diuretics, ultrafiltration, or equivalent) and overnight stay
Time Frame: From date of randomization to date of event, assessed for a minimum of 24 months and up to 60 months
Arm/Group | CRT-P ON | CRT-P OFF
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Quality of Life (QoL)
Description: The quality of life between study groups and the change in quality of life over time between study groups using clinically accepted quality of life measures.
  Note: No subjects completed 24 months of follow-up, so this objective could not be analyzed.
  Two QOL questionnaires were used in the study.
  EQ-5D: scores typically range from 0-1, where higher scores reflect better quality of life KCCQ: scores range from 0-100, where higher scores reflect better quality of life
Time Frame: Assessed from baseline visit to 24-month follow-up visit
Arm/Group | CRT-P ON | CRT-P OFF
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Reverse Remodeling by Echocardiography
Description: The change in LVEF between study groups.
  Note: No subjects completed 24 months of follow-up, so this objective could not be analyzed.
Time Frame: Assessed from baseline visit to 24-month follow-up visit
Arm/Group | CRT-P ON | CRT-P OFF
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the point of enrollment. Due to the study being halted early, no subject was followed for more than 14 months post-implantation of a CRT device.
Groups:
- CRT-P OFF: Subjects who were implanted with a CRT-P device and device programmed to minimal pacing at 40 beats/minute. Device and arrhythmia diagnostics may remain enabled.
Arm/Group | No Implant Attempt | CRT-P ON | CRT-P OFF
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/19 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/18 | 1/19 | 2/7
Other Adverse Events (participants affected / at risk) | 0/18 | 6/19 | 2/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | No Implant Attempt (N=18) | CRT-P ON (N=19) | CRT-P OFF (N=7)
Atrial flutter (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Device dislocation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) — Lead dislodgement
Enterocolitis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Metabolic encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | No Implant Attempt (N=18) | CRT-P ON (N=19) | CRT-P OFF (N=7)
Device dislocation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Ischaemic cardiomyopathy (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Wound infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Implant site haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No